CLINICAL TRIAL: NCT05419453
Title: Microbiome Composition and Function Contributes to Cognitive Impairment and Neuroinflammation in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: California State University, San Bernardino (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Jacob Jones, Clinical Psychologist, California State University, San Bernardino
Other Study IDs: SC3NS124906 (NIH)
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Cognition
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood, fecal matter
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's: Those with Parkinson's Disease

SUMMARY:
Cognitive impairment is a common non-motor symptom among individuals living with Parkinson's disease (PD). Traditionally, cognitive impairment is thought to reflect disruptions in dopaminergic frontal-striatal systems. However, the current conceptualization does not thoroughly explain the heterogeneous profiles or trajectories of cognitive impairment in PD; suggesting that alternative mechanisms may contribute to cognitive impairments. Identification of alternative mechanisms of cognitive impairment may lead to better prognostic prediction and yield novel treatment targets. The gut is implicated as a site of early pathology in PD. Early signs of PD pathology (alpha synuclein and Lewy body aggregates) are detected in the gastrointestinal tract years before motor symptoms manifest. Recent studies provide evidence that individuals with PD have an altered gut-bacterial composition (termed dysbiosis) relative to controls. To date, dysbiosis is linked to more severe motor symptoms and certain non-motor symptoms (constipation, REM behavioral sleep disorder) in PD, but the relationship between dysbiosis and cognitive impairment remains unknown. Animal studies support the hypothesis that microbiota composition play a direct role in cognitive impairment. Germ free (GF) mice demonstrate deficits in cognition. Specifically, findings suggest that a disrupted gut- microbial environment in conjunction with elevated stress hormones may create an imbalance of pro- inflammatory vs. anti-inflammatory cytokines that induces potentially reversible cognitive impairments. In human studies among individuals with PD, neuroinflammatory markers are associated with cognitive impairment. However, the relationship between dysbiosis, neural inflammation and cognitive functioning remains unknown. This model has incredible clinical implications, as microbiota dysbiosis may represent a reversible risk factor for cognitive impairment. The proposed study will examine the hypothesis that dysbiosis contributes to increased neuroinflammation and cognitive impairment. Microbiota composition/function, neuroinflammatory markers and cognitive functioning will be examined in 100 participants with PD. Analyses of microbiota composition/function will examine abundance of amplicon sequence variants (ASVs; 16s), bacterial species/strains (metagenomics), microbial genes, and functional pathways. The investigators hypothesize that microbiota composition/function will be associated with inflammatory markers (e.g. interleukin-6, tumor necrosis factor-alpha, c-reactive protein) and cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease

Exclusion Criteria:

* Use of antibiotics or immunosuppressant medications within the last 3 months, history of psychiatric hospitalizations, stroke, epilepsy, head injury resulting in a loss of consciousness for more than 30 minutes, Alzheimer's disease or other significant brain injury or neurologic event, history of inflammatory gastrointestinal diseases such as Crohn's, Celiac's disease or irritable bowel syndrome

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Cognitive Impairment | 4 hours
  Cognitive functioning as measured by a composite measure (average) of all neuropsychological tests

CONTACTS AND LOCATIONS:
Locations (1):
- California State University San Bernardino, San Bernardino, California, United States